CLINICAL TRIAL: NCT03116698
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Study to Evaluate the Dose-Response Relationship of the Efficacy and Safety of Two Concentrations of DFD-07 Cream, in Subjects With Actinic Keratosis (AK) of the Face and/or Scalp Over a 12-week Treatment Period.
Brief Title: A Study to Evaluate Two Concentrations of DFD-07 Cream, in Subjects With Actinic Keratosis (AK) of the Face and/or Scalp Over a 12-week Treatment Period
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFD-07-CD-002
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose DFD07 once daily (Experimental)
  Interventions: Drug: Low dose DFD07 once daily
- High dose DFD07 once daily (Experimental)
  Interventions: Drug: High dose DFD07 once daily
- High dose DFD07 twice daily (Experimental)
  Interventions: Drug: High dose DFD07 twice daily
- Placebo twice daily (Placebo Comparator)
  Interventions: Drug: Placebo twice daily

INTERVENTIONS:
Drug: Low dose DFD07 once daily — Low dose DFD07 once daily
  Arms: Low dose DFD07 once daily
Drug: High dose DFD07 once daily — High dose DFD07 once daily
  Arms: High dose DFD07 once daily
Drug: High dose DFD07 twice daily — High dose DFD07 twice daily
  Arms: High dose DFD07 twice daily
Drug: Placebo twice daily — Placebo twice daily
  Arms: Placebo twice daily

SUMMARY:
Once or twice daily 12 week treatment in patients with Actinic Keratosis randomized to treatment in one of four arms.

ELIGIBILITY:
Inclusion:

1. Subject understands the study procedures, is willing to comply with the study procedures and required visits, and agrees to participate by giving written informed consent. Subjects with a legal guardian, must have the written informed consent of the legal guardian.
2. Subject (or legal guardian) must be willing to authorize use and disclosure of protected health information collected for the study.
3. Subjects must have 5 or more AK lesions that are non-hypertrophic and non-hyperkeratotic, contained within a single contiguous approximately 5 cm x 5 cm (25 cm2) region of face and/or scalp.
4. Subjects must be 18 years of age or older. Male and female subjects can be enrolled.
5. Female subjects of childbearing potential must agree to use contraception during the study which can include abstinence with an adequate secondary option should the subject become sexually active. All women of childbearing potential must complete a urine pregnancy test at the Baseline Visit (Visit 2) and the test result must be negative to be eligible for enrollment.

   A female is considered of childbearing potential unless she is:
   1. postmenopausal for at least 12 months prior to study product administration;
   2. without a uterus and/or both ovaries; or has been surgically sterile (i.e., tubal ligation) for at least 6 months prior to study product administration.

   Reliable methods of contraception are:
   1. hormonal methods or intrauterine device in use more than 90 days prior to study product administration; or
   2. barrier methods plus spermicide in use at least 14 days prior to study product administration.
   3. partner has had a vasectomy at least 3 months previous to study product administration.
   4. Essure

   Exception: Sexually inactive female subjects of childbearing potential are not required to practice a reliable method of contraception and may be enrolled at the investigator's discretion provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study. An abstinent female must agree that if she becomes sexually active during the study she will use an acceptable form of contraception.
6. Subjects must agree not to use any product on the treatment area during the entire course of study except for Investigator-approved cleanser, sunscreen, wash, and non-medicated make-up. Subjects should continue to use these Investigator-approved products for the duration of the study and should avoid any changes in these consumer products.
7. Subjects must be willing to comply with sun avoidance measures for the face including use of Investigator-approved sunscreen and/or hats, have limited sun exposure time, and have no tanning bed use.
8. Subjects must be in good general health as determined by the Investigator and supported by the medical history, and normal or not clinically significant abnormal vital signs (blood pressure and pulse rate). Subjects are eligible if:

   * Systolic blood pressure (BP) < 160 and > 85 mmHg
   * Diastolic BP < 100 and > 50 mmHg

Exclusion:

1. Known or suspected hypersensitivity to any non-steroidal anti-inflammatory drugs (NSAID) or any component of the formulation of the study medication, including a history of asthma, urticarial, or other allergic-type reactions after taking aspirin or other NSAIDs.
2. Known or suspected allergy to sulfonamides.
3. Clinical evidence of severe, uncontrolled autoimmune, cardiovascular, gastrointestinal, hematological, hepatic, neurologic, pulmonary or renal disease.
4. Recent (within 6 months) or planned coronary artery bypass graft surgery.
5. Significant history (within the past year) of alcohol or drug abuse.
6. Participation in any clinical research study within 30 days of the Baseline Visit.
7. Concomitant use of cosmetics or other topical drug products on or near the selected treatment area, except for Investigator-approved cleanser, sunscreen, wash, and non-medicated makeup.
8. Cosmetic or therapeutic procedures (e.g. laser, peeling, photodynamic therapy) within 2 weeks and within 2 cm of the selected treatment area.
9. Other skin conditions within the selected treatment area (e.g. rosacea, psoriasis, atopic dermatitis, eczema, basal or squamous cell carcinoma or albinism).
10. Any systemic cancer therapy or diagnosis within 6 months of the Baseline Visit.
11. Females who are pregnant or lactating or planning to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R. Sidgiddi, M.D., Study Director — Dr. Reddy's Laboratories
Locations (20):
- United States (20):
  - Investigator Site 3, Cerritos, California
  - Investigator Site 1, Fremont, California
  - Investigator Site 9, Palm Springs, California
  - Investigator Site 18, Santa Ana, California
  - Investigator Site 16, Boca Raton, Florida
  - Investigator Site 8, Lake City, Florida
  - Investigator Site 7, Miami, Florida
  - Investigator Site 19, Miami, Florida
  - Investigator Site 20, Miami Lakes, Florida
  - Investigator Site 17, Ormond Beach, Florida
  - Investigator Site 6, West Palm Beach, Florida
  - Investigator Site 13, Verona, New Jersey
  - Investigator Site 15, Stony Brook, New York
  - Investigator Site 14, Fort Washington, Pennsylvania
  - Investigator Site 10, Austin, Texas
  - Investigator Site 4, Houston, Texas
  - Investigator Site 5, Plano, Texas
  - Investigator Site 11, San Antonio, Texas
  - Investigator Site 2, San Antonio, Texas
  - Investigator Site 12, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 240 subjects were expected to be randomized, but 238 subjects were randomized and included in the ITT population and 183 subjects were included in the Per Protocol population.
Groups:
- DFD07 - 1.25% Once Daily: Low dose DFD07 (1.25%) once daily:
  The active investigational product was applied once daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. The dose for the study product was a maximum of 0.5 g per application to the entire 5 cm x 5 cm area on the face and/or scalp for a maximum dose of 0.5 g per day. In this group, the randomized active DFD-07 (celecoxib) Cream product was applied once daily in the evening, while the Vehicle for DFD-07 Cream was applied once daily in the morning to keep the blinding between groups.
- DFD07 - 2.5% Once Daily: High dose DFD07 (2.5%) once daily:
  The active investigational product was applied once daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. The dose for the study product was a maximum of 0.5 g per application to the entire 5 cm x 5 cm area on the face and/or scalp for a maximum dose of 0.5 g per day. In this group, the randomized active DFD-07 (celecoxib) Cream product was applied once daily in the evening, while the Vehicle for DFD-07 Cream was applied once daily in the morning to keep the blinding between groups.
- DFD07 - 2.5% Twice Daily: High dose DFD07 (2.5%) twice daily: The active investigational product was applied twice daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. The dose for the study product was a maximum of 0.5 g per application to the entire 5 cm x 5 cm area on the face and/or scalp for a maximum dose of 1.0 g per day.
- Vehicle Twice Daily: Vehicle twice daily:
  The Vehicle product was applied twice daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. The dose for the Vehicle product was a maximum of 0.5 g per application to the entire 5 cm x 5 cm area on the face and/or scalp for a maximum dose of 1.0 g per day.
Period: Overall Study
Arm/Group | DFD07 - 1.25% Once Daily | DFD07 - 2.5% Once Daily | DFD07 - 2.5% Twice Daily | Vehicle Twice Daily
Started | 62 | 57 | 62 | 57
Completed | 56 | 51 | 54 | 55
Not Completed | 6 | 6 | 8 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 5 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- DFD07 Cream 1.25% Once Daily: DFD07 Cream (celecoxib 1.25%) once daily:
  The active investigational product was applied once daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. In this group, the randomized active DFD-07 (celecoxib 1.25%) Cream product was applied once daily in the evening, while the Vehicle for DFD-07 Cream was applied once daily in the morning to keep the blinding between groups.
- DFD07 Cream 2.5% Once Daily: DFD07 Cream (celecoxib 2.5%) once daily:
  The active investigational product was applied once daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment. In this group, the randomized active DFD-07 (celecoxib 2.5%) Cream product was applied once daily in the evening, while the Vehicle for DFD-07 Cream was applied once daily in the morning to keep the blinding between groups.
- DFD07 Cream 2.5% Twice Daily: DFD07 Cream (celecoxib 2.5%) twice daily:
  The active investigational product was applied twice daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment.
- Vehicle Cream Twice Daily: Vehicle Cream (celecoxib 0%) twice daily:
  The Vehicle Cream was applied twice daily for 12 weeks to cover the entire lesional area (5 cm x 5 cm) on the face and/or scalp identified by the Investigator for treatment.
- Total: Total of all reporting groups
Arm/Group | DFD07 Cream 1.25% Once Daily | DFD07 Cream 2.5% Once Daily | DFD07 Cream 2.5% Twice Daily | Vehicle Cream Twice Daily | Total
Number analyzed (Participants) | 62 | 57 | 62 | 57 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.74 (11.00) | 65.71 (11.54) | 69.74 (11.60) | 66.66 (11.21) | 67.71 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 23 | 22 | 90
  Male | 37 | 37 | 39 | 35 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 18 | 17 | 66
  Not Hispanic or Latino | 46 | 42 | 43 | 38 | 169
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 1 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 58 | 54 | 61 | 54 | 227
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 57 | 62 | 57 | 238

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Complete Clearance of AK Lesions at the End of Study Visit at 16 Weeks
Description: The proportion of subjects with complete clearance (absence of clinically visible or palpable AK lesions in the treatment area) of AK lesions at the End of Study Visit at 16 weeks (12 weeks treatment and 4 weeks treatment-free follow-up)
Time Frame: 16 Weeks
Population: Intent To Treat (ITT) population defined as all subjects who were randomized and dispensed study medication.
Measure: Count of Participants; unit: Participants
Groups:
- DFD07 Cream (Celecoxib 1.25%) Once Daily: DFD07 Cream (Celecoxib 1.25%) Once daily for 12 weeks followed by 4 weeks treatment-free period. In this group active treatment was applied once daily in the evening and Vehicle treatment was applied once daily in the morning for 12 weeks to maintain study blind.
- DFD07 Cream (Celecoxib 2.5%) Once Daily: DFD07 Cream (Celecoxib 2.5%) Once daily for 12 weeks followed by 4 weeks treatment-free period. In this group active treatment was applied once daily in the evening and Vehicle treatment was applied once daily in the morning for 12 weeks to maintain study blind.
- DFD07 Cream (Celecoxib 2.5%) Twice Daily: DFD07 Cream (Celecoxib 2.5%) Twice daily for 12 weeks followed by 4 weeks treatment-free period
- Vehicle Cream (Celecoxib 0%) Twice Daily: Vehicle Cream (Celecoxib 0%) Twice daily for 12 weeks followed by 4 weeks treatment-free period
Arm/Group | DFD07 Cream (Celecoxib 1.25%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Twice Daily | Vehicle Cream (Celecoxib 0%) Twice Daily
Number analyzed (Participants) | 62 | 57 | 62 | 57
Participants | 6 | 9 | 10 | 7

2. Secondary Outcome: Proportion of Subjects With Partial Clearance at Week 16
Description: Proportion of subjects with partial clearance of AK lesions at week 16 (12 weeks treatment and 4 weeks treatment free follow up period)
Time Frame: 16 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | DFD07 Cream (Celecoxib 1.25%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Twice Daily | Vehicle Cream (Celecoxib 0%) Twice Daily
Number analyzed (Participants) | 62 | 57 | 62 | 57
Participants | 14 | 19 | 17 | 18

ADVERSE EVENTS:
Time Frame: All Adverse events that occurred during the treatment period from the Baseline visit (Day 1) until the end of study (Week 16)
Arm/Group | DFD07 Cream (Celecoxib 1.25%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Once Daily | DFD07 Cream (Celecoxib 2.5%) Twice Daily | Vehicle Cream (Celecoxib 0%) Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/57 | 2/62 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/57 | 2/62 | 0/57
Other Adverse Events (participants affected / at risk) | 18/62 | 8/57 | 21/62 | 11/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD07 Cream (Celecoxib 1.25%) Once Daily (N=62) | DFD07 Cream (Celecoxib 2.5%) Once Daily (N=57) | DFD07 Cream (Celecoxib 2.5%) Twice Daily (N=62) | Vehicle Cream (Celecoxib 0%) Twice Daily (N=57)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject died due to cardiovascular disease 23 days after the last study drug application, prior to completing end-of-study procedures. The subject was in the DFD-07 Cream, 2.5% BID group. The Investigator determined it to be unrelated to study drug
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject passed out and died at home five days after last study drug application. Autopsy was not performed but the cause of death was reported as COPD. The Investigator determined the death to be unrelated to the study drug,
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DFD07 Cream (Celecoxib 1.25%) Once Daily (N=62) | DFD07 Cream (Celecoxib 2.5%) Once Daily (N=57) | DFD07 Cream (Celecoxib 2.5%) Twice Daily (N=62) | Vehicle Cream (Celecoxib 0%) Twice Daily (N=57)
Infections (Infections and infestations) | 7 | 2 | 5 | 2
Cardiac Disorders (Cardiac disorders) | 0 | 0 | 1 | 1
Gastrointestinal Disorders (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Application site events (General disorders) | 1 | 0 | 1 | 1
Immune disorders (Immune system disorders) | 1 | 0 | 0 | 2
Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Laboratory test abnormalities (Investigations) | 1 | 1 | 0 | 1
Metabolic disorders (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Nervous system disorders (Nervous system disorders) | 2 | 2 | 3 | 1
Respiratory events (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Skin disorders (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 2
Procedures (Surgical and medical procedures) | 2 | 0 | 0 | 1
Vascular disorders (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03116698/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03116698/SAP_001.pdf